CLINICAL TRIAL: NCT05892185
Title: A Randomized, Single-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Glaucoma Implant in Primary Open Angle Glaucoma.
Brief Title: Evaluate the Efficacy and Safety of Glaucoma Implant in Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mingche Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC-001-081
Record Dates: First submitted 2023-05-23; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma
Keywords: Glaucoma Implant
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GELA (Experimental): Participants underwent at least one preoperative visit and had GELA implantation on Day 0 (The day of surgery)
  Interventions: Device: GELA
- XEN (Active Comparator): Participants underwent at least one preoperative visit and had XEN gel stent implantation on Day 0 (The day of surgery).
  Interventions: Device: XEN

INTERVENTIONS:
Device: GELA — GELA glaucoma implant
  Arms: GELA
Device: XEN — XEN gel stent implant
  Arms: XEN

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of glaucoma device in the treatment of primary open-angle glaucoma.

DETAILED DESCRIPTION:
A prospective, randomized, single-blind, positive control design was used to study primary open-angle glaucoma. Eligible subjects were screened and randomly assigned to the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria

* Patients with a clinical diagnosis of primary open-angle glaucoma (POAG) who could undergo minimally invasive glaucoma surgery (MIGS) as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2024-01-12 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
Success rate at 6 months after surgery | 6 months
  Success rate defined as the percentage of total cases in which IOP decreased ≥20% and/or IOP ≤21mmHg while using the same or lower amount of IOP-lowering medications compared to baseline at 6 month after surgery.

SECONDARY OUTCOMES:
IOP reduction | 6 months
  The IOP of the subjects before and 6 months after surgery was calculated in both experiment group and control group.
topical IOP-lowering medications | 6 months
  Counting by class of drug of topical IOP lowering medications before and 6-month after surgery.
Success rate 12 months after operation | 12 months
  Success rate defined as the percentage of total cases in which IOP decreased ≥20% and/or IOP ≤21mmHg while using the same or lower amount of IOP-lowering medications compared to baseline at 12 month after surgery.
Adverse event | 12 months
  Adverse events was recorded and summarized.

IPD SHARING:
Plan to Share IPD: No